CLINICAL TRIAL: NCT00110955
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Darbepoetin Alfa for the Treatment of Anemia in Subjects With Non-Myeloid Malignancy Receiving Multicycle Chemotherapy
Brief Title: Treatment of Anemia in Subjects With Non-Myeloid Malignancy Receiving Multicycle Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20030232
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Anemia; Non-Myeloid Malignancies
Keywords: Non-myeloid malignancy; Chemotherapy-induced anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Darbepoetin alfa - Group A (Experimental)
  Interventions: Drug: Darbepoetin alfa
- Placebo- Group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa — Q3W 300 mcg darbepoetin alfa
  Arms: Darbepoetin alfa - Group A
Drug: Placebo — Q3W dosing of placebo
  Arms: Placebo- Group B

SUMMARY:
The purpose of this study is to compare the effect of darbepoetin alfa against placebo for the treatment of anemia in subjects with non-myeloid malignancies receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with non-myeloid malignancy
* At least 12 additional weeks of cyclic cytotoxic chemotherapy anticipated regardless of schedule
* Hemoglobin concentration less than 11.0 g/dL within 24 hours before randomization
* Adequate serum folate and vitamin B12
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Of legal age at the time written informed consent is obtained

Exclusion Criteria:

* Known history of seizure disorder
* Known primary hematologic disorder causing anemia other than non-myeloid malignancies
* Unstable/uncontrolled cardiac condition
* Clinically significant inflammatory disease
* Other diagnoses not related to the cancer which can cause anemia
* Inadequate renal and liver function
* Iron deficiency
* Known positive test for HIV infection
* Previously suspected of or confirmed to have neutralizing antibodies to rHuEPO
* Received more than 2 red blood cell (RBC) transfusions within 4 weeks of randomization; or any RBC transfusion within 14 days before randomization; or any planned RBC transfusion between randomization and study day 1
* Received any erythropoietic therapy within 4 weeks of study day 1 or any planned erythropoietic therapy between randomization and study day 1
* Other investigational procedures
* Currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject receiving other investigational agent(s)
* Pregnant or breast feeding
* Not using adequate contraceptive precautions
* Previously randomized into this study
* Known hypersensitivity to any products to be administered
* Concerns for subject's compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2004-02; Primary Completion 2005-03 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Incidence of red blood cell (RBC) transfusion from week 5 to End of Treatment Period (EOTP) | from week 5 to EOTP

SECONDARY OUTCOMES:
Incidence of achieving a hemoglobin concentration of greater than or equal to 11 g/dL in the absence of RBC transfusions in the preceding 28 days from week 5 to EOTP | from week 5 to EOTP
Number of RBC transfusions from week 5 to EOTP | from week 5 to EOTP
Change in FACT-Fatigue subscale score from baseline to EOTP | from baseline to EOTP
Change in FACT-G Physical Well-being subscale from baseline to EOTP | from baseline to EOTP
Incidence and severity of adverse events | throughout study
Incidence of hemoglobin concentration greater than 13.0 g/dL at any time on study | at any time on study
Change in FACT-G total score from baseline to EOTP | from baseline to EOTP
Incidence of an increase in hemoglobin concentration greater than or equal to 2 g/dL in a 28-day window and any negative clinical consequences | throughout study
Change in EQ-5D Thermometer from baseline to EOTP | from baseline to EOTP
Change in BSI Anxiety scale score from baseline to EOTP | from baseline to EOTP
Change in BSI Depression scale score from baseline to EOTP | from baseline to EOTP
Change in number of caregiver hours from baseline to EOTP | from baseline to EOTP
Incidence of a confirmed antibody formation to darbepoetin alfa | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Hernandez E, Ganly P, Charu V, Dibenedetto J, Tomita D, Lillie T, Taylor K; ARANESP 20030232 Study Group. Randomized, double-blind, placebo-controlled trial of every-3-week darbepoetin alfa 300 micrograms for treatment of chemotherapy-induced anemia. Curr Med Res Opin. 2009 Sep;25(9):2109-20. doi: 10.1185/03007990903084164. PMID 19601709
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20030232_Posting_Summ_NESP.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/